CLINICAL TRIAL: NCT02444351
Title: Botulinum Toxin Type A Injection Into the Gastrocnemius Muscle for Treatment of Nocturnal Calf Cramps in Patients With Lumbar Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2015-0169
Record Dates: First submitted 2015-04-28; First posted 2015-05-14 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2017-01

CONDITIONS: Spinal Stenosis With Nocturnal Calf Cramps
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Other: no intervention
- botox group (Experimental)
  Interventions: Drug: botulinum toxin type A (Nabota®) injection into the gastrocnemius muscle

INTERVENTIONS:
Drug: botulinum toxin type A (Nabota®) injection into the gastrocnemius muscle — ultrasound-guided botulinum toxin type A (Nabota®, Daewoong co. Seoul, Korea) injection into the gastrocnemius muscle (maximum 200unit per each calf).
  Arms: botox group
Other: no intervention — Patients in the control group will not receive any injection on the gastrocnemius muscle.
  Arms: control group

SUMMARY:
Nocturnal calf cramps is a common complaint in patients with lumbar spinal stenosis. The purpose of this study is to evaluate the effect of botulinum toxin A injection into the gastrocnemius muscle in lumbar spinal stenosis patients receiving conservative therapy. We will compare pain score, insomnia severity, functional ability, patient satisfaction, and neurophysiological variables change using electrical stimulator between control (conservative management for spinal stenosis) and botox group (conservative management for spinal stenosis plus botox injection into the gastrocnemius muscle).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed lumbar spinal stenosis with MRI finding
2. nocturnal calf cramps symptoms at least once per week

Exclusion Criteria:

1. electrolyte disorder
2. congenital muscle disease
3. muscle cramps related medication (statins, diuretics, calcium channel blockers, anticonvulsants etc.)
4. cognitive impairments

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Pain score | follow up 2 weeks (14 days) after injection
  A comparison of pain score between control (conservative management for spinal stenosis) and botox group (conservative management for spinal stenosis plus botox injection into the gastrocnemius muscle).

SECONDARY OUTCOMES:
patient satisfaction questionnaire using 0 to 4 scale | follow up 3 months after injection
  assessment of patient satisfaction using 0 to 4 scale (0; very dissatisfied, 1; dissatisfied, 2; fair, 3; satisfied, 4; very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park SJ, Yoon KB, Yoon DM, Kim SH. Botulinum Toxin Treatment for Nocturnal Calf Cramps in Patients With Lumbar Spinal Stenosis: A Randomized Clinical Trial. Arch Phys Med Rehabil. 2017 May;98(5):957-963. doi: 10.1016/j.apmr.2017.01.017. Epub 2017 Feb 14. PMID 28209505